CLINICAL TRIAL: NCT04596904
Title: The Effect of Lavender Smell on Anxiety Due to Endoscopic Procedures
Brief Title: The Effect of Lavender Smell on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fatmanur Ince Ozgenel, Nurse, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8680
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Clinical research with herbal products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender oil group (Experimental): Individuals, for 10 days, 3 drops of cotton drops of lavender oil, put on the shoulder parts, between 21:00 and 21:05 will smell every evening.
  Interventions: Other: Lavender oil application group
- Distilled water group (Placebo Comparator): Individuals, for 10 days, 3 drops of cotton drops of distilled water, put on the shoulder parts, between 21:00 and 21:05 will smell every evening.
  Interventions: Other: Distilled water application group

INTERVENTIONS:
Other: Lavender oil application group — Individuals, for 10 days, 3 drops of cotton drops of lavender oil, put on the shoulder parts, between 21:00 and 21:05 will smell every evening.
  Arms: Lavender oil group
Other: Distilled water application group — Individuals, for 10 days, 3 drops of cotton drops of distilled water, put on the shoulder parts, between 21:00 and 21:05 will smell every evening.
  Arms: Distilled water group

SUMMARY:
Esophagogastroduodenoscopy and colonoscopy are invasive procedures that enable the diagnosis, diagnosis, treatment, biopsy, photo and video recording of the gastrointestinal tract. It has an important place in clinical use for diagnosis and treatment and these procedures are common. When the studies are examined; while the prevalence of gastroesophageal reflux disease was 8.8% -25.9% in Europe, approximately 20% of the population in the world were found to have dyspeptic complaints. In the UK, 41,000 new colorectal cancers were diagnosed in 2014 and 132700 new cases were detected in the United States in 2015. In the European Union countries, the incidence of gastrointestinal cancer reported in 2012 is 684,000 cases.

During endoscopic interventions in our country; in Turkey; people may experience high levels of anxiety considering the negative consequences of discomfort and pain.In such cases, nurses should make attempts to reduce the anxiety of the person by predicting that people may have anxiety. Non-pharmacological methods that may reduce anxiety include; pre-treatment training, aromatherapy, acupuncture, hypnosis. Eliminating or reducing anxiety as much as possible will help increase the comfort of both the patient and the endoscopist in these invasive procedures. In our study, our aim was to evaluate the effect of non-pharmacological methods on the preoperative lavender smell.

DETAILED DESCRIPTION:
Type and purpose of the study: This randomized controlled trial was planned to evaluate the effect of volatile lavender oil on the level of instantaneous and sustained anxiety level of the patients undergoing endoscopic procedure.

Time and place of study:

The research is carried out in Eskişehir Osmangazi University Gastroenterology Polyclinic.

Universe and sample: The population of the study was applied to the gastroenterology outpatient clinic for diagnosis and diagnosis. The sample of the research sample will be composed of people who meet the sample selection criteria in the specified universe.Chi-Square Test Power analysis was used to determine the sample number of the study. The statistical power was calculated as 118 people with 82%, alpha 0.05, beta 0,1741 errors and 59 persons in group A and 59 persons in group B. In the calculation of the power analysis, Hu et al. (2010) evaluated the effect of lavender in the management of anxiety related to colonoscopy.

Randomization: Within the scope of the study, written consent was obtained after the individuals were informed by the researchers. Randomization method was randomized to two groups [(lavender oil group (A), control group (B)]. The registration numbers and the group numbers of the individuals will be delivered to the researchers in a closed envelope and the lavender oil / distilled water will be sniffed according to the group of the individual before the procedure.

There are differences in the level of anxiety related to esophagogastroduodenoscopy and colonoscopy. For this reason, randomization of the patients to groups will be tried to be matched with the case of esophageogudroduodenoscopy and colonoscopy. Patients in the same group of patients will also be included in group B according to the type of procedure in each group (esophagogastroduodenoscopy / colonoscopy).

Preparation of aromatic oils: In the light of the information obtained from the studies evaluating the effect of lavender oil on anxiety, lavender oil with a sedative effect was used in one group, while the other group was determined to use jojoba, sunflower, jasmine, rosemary, grape seed, tea tree oils without sedative effect.

Lavender oil (Lavandula hybrida): The volatile lavender oil to be used for the enterprise will be taken from a reliable plant product company and the company has got the operation registration and TS EN ISO 9001: 2008 quality certificates from the Ministry of Food, Agriculture and Livestock by G06-3231. After 10 days of 3 drops of lavender oil on the cotton pad, the prepared cotton pad will be placed on the shoulder dress. Application and evaluation: The data of the study will be collected in the first and second stage in a total of 2 weeks; First stage:Individual presentation form, State Trait Anxiety Inventory-I, II will be applied to the individuals who have been given an appointment to perform esophagogastroduodenoscopy and colonoscopy in the gastroenterology outpatient clinic, then A and B group individuals will be informed by the healthcare professional about the application of lavender oil / distilled water at home. For 10 days at home, group A patients receive lavender oil; Group B patients will smell distilled water every evening between 21.00-21.05 for 5 minutes.

Second stage: State Trait Anxiety Inventory-I, II will be filled before sedation in patients coming to the outpatient clinic for esophagogastroduodenoscopy and colonoscopy, vital signs (heart rate, respiratory rate, blood pressure arterial) to be evaluated and the sedation protocol prescribed by the physician. No changes shall be made to the screening, diagnosis and treatment of individuals during the trial.

Individual presentation form: Socio-demographic characteristics of patients (age, gender, educational status, marital status, information to support the patient's care) and disease-related features (diagnosis, treatment, duration of disease) is a form of questions about.

State Trait Anxiety Inventory (I, II) is a self-assessment questionnaire consisting of short expressions. This is a Likert-type scale, a four-degree scale ranging from None "to" Completely. It includes the description of how an individual feels himself / herself in a certain moment and under certain conditions and taking into account his / her feelings about the situation he / she is in. Cronbach alpha internal consistency coefficients in reliability analysis;0.94-0.96 for State Anxiety Inventory, for The Trait Anxiety Inventory is between 0.83 and 0.87. There are two types of expressions in State-Trait Anxiety Inventories. Direct expressions express negative feelings and reversed expressions express positive feelings. In the State Anxiety Inventory, the terms reversed are 1,2,5,8,10,11,15,16,19 and 20 items. On the Trait Anxiety Inventory, the inverse statements constitute 21,26,27,30,33,36 and 39th items. After the total weight of the direct and inverted expressions are found, the total weight score of the reverse expressions is subtracted from the total weight score obtained for the direct expressions. A predetermined and unchanged value is added to this number. This constant value is 50 for the State Anxiety Inventory and is 35 for the Trait Anxiety Inventory. The recent value is an individual's anxiety score

ELIGIBILITY:
Inclusion Criteria: The volunteers who will undergo esophagogastroduodenoscopy or colonoscopy to the gastroenterology outpatient clinic were included in the study.

-

Exclusion Criteria: Having cardiovascular disease, Asthma Known history of allergy To be diagnosed psychiatric disease (anxiety / panic attack / depression) To take anxiolytic medication (such as benzodiazepines, selective serotonin reuptake inhibitors, To use products such as antiperspirant, perfume, spray containing any fragrance to the hair and body before the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change of the State-Trait Anxiety Inventory Scores | Before the endoscopic procedure - on endoscopic procedure day
  An individual identification form and the State-Trait Anxiety Inventory were used to collect the data.It is a self-assessment questionnaire consisting of short statements.It includes the feature of describing how the individual feels at a certain moment and under certain conditions and responding by taking into account their feelings about the situation. In reliability analysis, Cronbach alpha internal consistency coefficients; 0.94-0.96 for State Anxiety Inventory; it is between 0.83 and 0.87 for the Trait Anxiety Inventory.The unchanged value for the State Anxiety Inventory is 50 and 35 for the Trait Anxiety Inventory. The last obtained value is the individual's anxiety score.

CONTACTS AND LOCATIONS:
Overall Officials: Fatmanur Ozgenel, Nurse, Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Fatmanur Ince Ozgenel, Eskişehir, Turkey (Türkiye)